CLINICAL TRIAL: NCT07349004
Title: Association Between PFO and Migraine With Aura: A Case-Control Observational Study With Genetic and Neurosonological Analysis
Brief Title: Neurogenetic And Hemodynamic Of Migraine Aura And Pfo
Acronym: PFOCUS
Status: Recruiting | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: PFOCUS
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Migraine With Aura
Keywords: patent foramen ovale; migraine with aura; CADASIL
MeSH Terms: conditions — Migraine with Aura; Foramen Ovale, Patent; CADASIL | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Patients with migraine with aura who have a patent foramen ovale (MAPFO+)
  Interventions: Other: Intervention
- Arm 2: Patients with migraine with aura without patent foramen ovale (MAPFO-)
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Neurosonological protocol with continuous Doppler monitoring for microemboli detection, cerebrovascular reactivity and dynamic cerebral autoregulation testing, and a contrast-enhanced shunt study using agitated saline; blood samples for whole-exome sequencing and platelet aggregation studies.

SUMMARY:
The PFOCUS Study aims to clarify the relationship between patent foramen ovale (PFO) and migraine with aura (MA). Patients diagnosed with MA according to ICHD-3 criteria will be classified as cases (PFO+) or controls (PFO-) based on the presence or absence of a right-to-left shunt detected by transcranial Doppler or a previously documented PFO. The study will enroll 240 adult participants over 36 months.

The primary objective is to determine whether genetic variants differ significantly between patients with MA with and without PFO. Secondary objectives include assessing cerebral blood flow regulation and platelet function in patients with MA with and without PFO.

Participants will undergo a single study visit including the collection of demographic and clinical data and a comprehensive neurosonological assessment. This will include microembolic signal counts, cerebrovascular reactivity testing, and a contrast-enhanced transcranial Doppler study for shunt detection. Blood samples will be collected for whole-exome sequencing (with a focus on NOTCH3 and an expanded gene panel) and for platelet aggregometry.

The study is expected to provide new insights into the biological mechanisms linking PFO and MA-potentially involving endothelial dysfunction, altered vascular smooth muscle responses, or platelet activation-thereby informing prevention strategies and guiding future research.

DETAILED DESCRIPTION:
The PFOCUS study is a prospective, case-control observational investigation designed to explore the biological, vascular, and genetic factors associated with the coexistence of migraine with aura (MA) and patent foramen ovale (PFO). Epidemiological evidence indicates that individuals with MA have an increased risk of ischemic stroke even in the absence of traditional vascular risk factors. In parallel, a higher prevalence of PFO has been consistently reported in patients with MA, suggesting a potential role of PFO as a modifier of cerebrovascular risk. The mechanisms underlying this association are not fully understood and may involve factors beyond paradoxical embolism, including vascular dysfunction, altered cerebral hemodynamics, platelet activation, and genetic susceptibility.

The primary objective of the study is to compare the distribution of NOTCH3 gene variants and single nucleotide polymorphisms (SNPs) between patients with MA and PFO (PFO+) and patients with MA without PFO (PFO-). NOTCH3 encodes a receptor involved in vascular smooth muscle cell differentiation and small-vessel integrity, and pathogenic variants are known to cause cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL). Variants in this gene have also been associated with migraine phenotypes and alterations in cerebral small-vessel function. Given the role of NOTCH signaling pathways in cardiac septation and closure of the fetal foramen ovale, genetic variation in this pathway may contribute to both MA susceptibility and persistence of PFO.

Secondary objectives include: (1) assessing variants and SNPs in additional genes involved in NOTCH signaling, cardiac development, vascular regulation, and PFO heritability; (2) evaluating the relationship between genetic variants and the degree of right-to-left shunt; (3) comparing microembolic signals (MES) between PFO+ and PFO- participants using automated transcranial Doppler detection; (4) assessing cerebrovascular reactivity (CVR) and dynamic cerebral autoregulation (dCA) using standardized neurosonological protocols; and (5) comparing platelet function profiles between groups.

Each participant will undergo a single study visit. Data collection will include a structured clinical and demographic assessment, detailed characterization of migraine phenotype (including aura characteristics, attack frequency, and coexistence of migraine without aura), and review of available brain magnetic resonance imaging (MRI) findings when available. The neurosonological assessment will include continuous transcranial Doppler monitoring for MES detection, evaluation of CVR using breath-hold and hyperventilation maneuvers, and assessment of cerebral autoregulation using transfer function analysis, as well as contrast-enhanced detection of right-to-left shunt using agitated saline. Peripheral blood samples will be collected for genetic analysis and platelet function testing. Whole-exome sequencing will be performed, with subsequent analyses focused on a predefined panel of genes, including but not limited to NOTCH3, NOTCH1, JAG1, and HTRA1. Platelet aggregation studies will be conducted using standardized laboratory methods.

The planned sample size is 240 participants, equally distributed between the PFO+ and PFO- groups. This sample size is based on the expected prevalence of NOTCH3 SNPs and the anticipated between-group differences. Statistical analyses will include comparisons of allele and genotype frequencies, assessment of Hardy-Weinberg equilibrium, linkage disequilibrium analyses, and multivariable comparisons of neurosonological and platelet function parameters.

By integrating genetic, neurosonological, and hematological data, the PFOCUS study aims to characterize potential biological differences between patients with MA with and without PFO and to contribute to a better understanding of migraine-related vascular vulnerability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with aura (according to Chapter 1.2 of the International Classification of Headache Disorders, 3rd edition [ICHD-3])
* Age ≥ 18 years
* Both sexes
* Obtained written informed consent to participate in the study

Exclusion Criteria:

* History of congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of number of NOTCH3 genetic variants | T0 (day 1)
  To evaluate whether significant differences exist in the frequency of NOTCH3 genetic variants between patients with migraine with aura who have a patent foramen ovale (PFO+) and those without (PFO-). Min=0, max undefined.

SECONDARY OUTCOMES:
Comparison of number of genetic variants in other selected genes | T0 (day 1)
  To evaluate whether significant differences exist in the frequency of genetic variants in other selected genes between patients with migraine with aura who have a patent foramen ovale (PFO+) and those without (PFO-). Min=0, max undefined.
Correlation of genetic variants with shunt size | T0 (day 1)
  To assess whether the frequency of detected variants and SNPs correlates with the size of the right-to-left shunt in the PFO+ group (present vs absent).
Comparison in number of spontaneous microeboli | T0 (day 1)
  To evaluate differences in the number of cerebral microemboli between PFO+ and PFO- patients. Min=0, max undefined.
Comparison in cerebrovascular reactivity between PFO+ and PFO- patients | T0 (day 1)
  Evaluation of phase shift, gain and coherence for very low, low and high frequency obtained from Transfer function analysis (significant group difference: yes vs no)
Differences in platelet function profiles between PFO+ and PFO- patients | T0 (day 1)
  Evaluation of ASPI-test and ADP-test values obtained from Multiplate® analyzer (significant group difference: yes vs no)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Paolucci, Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna
Locations (1):
- IRCCS Istituto delle Scienze Neurologiche di Bologna - AUSL of Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West BH, Noureddin N, Mamzhi Y, Low CG, Coluzzi AC, Shih EJ, Gevorgyan Fleming R, Saver JL, Liebeskind DS, Charles A, Tobis JM. Frequency of Patent Foramen Ovale and Migraine in Patients With Cryptogenic Stroke. Stroke. 2018 May;49(5):1123-1128. doi: 10.1161/STROKEAHA.117.020160. Epub 2018 Apr 10. PMID 29636424
- [Background] Trabattoni D, Brambilla M, Canzano P, Becchetti A, Teruzzi G, Porro B, Fiorelli S, Muratori M, Tedesco CC, Veglia F, Montorsi P, Bartorelli AL, Tremoli E, Camera M. Migraine in Patients Undergoing PFO Closure: Characterization of a Platelet-Associated Pathophysiological Mechanism: The LEARNER Study. JACC Basic Transl Sci. 2022 Apr 13;7(6):525-540. doi: 10.1016/j.jacbts.2022.02.002. eCollection 2022 Jun. PMID 35818509
- [Background] Takagi H, Umemoto T; ALICE (All-Literature Investigation of Cardiovascular Evidence) Group. A meta-analysis of case-control studies of the association of migraine and patent foramen ovale. J Cardiol. 2016 Jun;67(6):493-503. doi: 10.1016/j.jjcc.2015.09.016. Epub 2015 Oct 31. PMID 26527111
- [Background] Schwaag S, Evers S, Schirmacher A, Stogbauer F, Ringelstein EB, Kuhlenbaumer G. Genetic variants of the NOTCH3 gene in migraine--a mutation analysis and association study. Cephalalgia. 2006 Feb;26(2):158-61. doi: 10.1111/j.1468-2982.2005.01007.x. PMID 16426270
- [Background] Schmidt H, Zeginigg M, Wiltgen M, Freudenberger P, Petrovic K, Cavalieri M, Gider P, Enzinger C, Fornage M, Debette S, Rotter JI, Ikram MA, Launer LJ, Schmidt R; CHARGE consortium Neurology working group. Genetic variants of the NOTCH3 gene in the elderly and magnetic resonance imaging correlates of age-related cerebral small vessel disease. Brain. 2011 Nov;134(Pt 11):3384-97. doi: 10.1093/brain/awr252. Epub 2011 Oct 17. PMID 22006983
- [Background] Rutten JW, Dauwerse HG, Gravesteijn G, van Belzen MJ, van der Grond J, Polke JM, Bernal-Quiros M, Lesnik Oberstein SA. Archetypal NOTCH3 mutations frequent in public exome: implications for CADASIL. Ann Clin Transl Neurol. 2016 Sep 28;3(11):844-853. doi: 10.1002/acn3.344. eCollection 2016 Nov. PMID 27844030
- [Background] Paolucci M, Vincenzi C, Romoli M, Amico G, Ceccherini I, Lattanzi S, Bersano A, Longoni M, Sacco S, Vernieri F, Pascarella R, Valzania F, Zedde M. The Genetic Landscape of Patent Foramen Ovale: A Systematic Review. Genes (Basel). 2021 Dec 6;12(12):1953. doi: 10.3390/genes12121953. PMID 34946902
- [Background] Paolucci M, Altamura C, Vernieri F. The Role of Endothelial Dysfunction in the Pathophysiology and Cerebrovascular Effects of Migraine: A Narrative Review. J Clin Neurol. 2021 Apr;17(2):164-175. doi: 10.3988/jcn.2021.17.2.164. PMID 33835736
- [Background] van Os HJA, Mulder IA, Broersen A, Algra A, van der Schaaf IC, Kappelle LJ, Velthuis BK, Terwindt GM, Schonewille WJ, Visser MC, Ferrari MD, van Walderveen MAA, Wermer MJH; DUST Investigators. Migraine and Cerebrovascular Atherosclerosis in Patients With Ischemic Stroke. Stroke. 2017 Jul;48(7):1973-1975. doi: 10.1161/STROKEAHA.116.016133. Epub 2017 May 19. PMID 28526767
- [Background] Menon S, Cox HC, Kuwahata M, Quinlan S, MacMillan JC, Haupt LM, Lea RA, Griffiths LR. Association of a Notch 3 gene polymorphism with migraine susceptibility. Cephalalgia. 2011 Feb;31(3):264-70. doi: 10.1177/0333102410381143. Epub 2010 Sep 2. PMID 20813781
- [Background] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Background] Li X, Xie L, Dai J, Zhou X, Chen T, Mao W. A whole-exome sequencing study of patent foramen ovale: investigating genetic variants and their association with cardiovascular disorders. Front Genet. 2024 May 14;15:1405307. doi: 10.3389/fgene.2024.1405307. eCollection 2024. PMID 38808331
- [Background] Lantz M, Sieurin J, Sjolander A, Waldenlind E, Sjostrand C, Wirdefeldt K. Migraine and risk of stroke: a national population-based twin study. Brain. 2017 Oct 1;140(10):2653-2662. doi: 10.1093/brain/awx223. PMID 28969391
- [Background] Kurth T, Chabriat H, Bousser MG. Migraine and stroke: a complex association with clinical implications. Lancet Neurol. 2012 Jan;11(1):92-100. doi: 10.1016/S1474-4422(11)70266-6. PMID 22172624
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Hu X, Zhou Y, Zhao H, Peng C. Migraine and the risk of stroke: an updated meta-analysis of prospective cohort studies. Neurol Sci. 2017 Jan;38(1):33-40. doi: 10.1007/s10072-016-2746-z. Epub 2016 Oct 26. PMID 27785579
- [Background] Hosseini-Alghaderi S, Baron M. Notch3 in Development, Health and Disease. Biomolecules. 2020 Mar 23;10(3):485. doi: 10.3390/biom10030485. PMID 32210034
- [Background] Guo ZN, Xing Y, Liu J, Wang S, Yan S, Jin H, Yang Y. Compromised dynamic cerebral autoregulation in patients with a right-to-left shunt: a potential mechanism of migraine and cryptogenic stroke. PLoS One. 2014 Aug 14;9(8):e104849. doi: 10.1371/journal.pone.0104849. eCollection 2014. PMID 25121485
- [Background] Dong B, Li Y, Ai F, Geng J, Tang T, Peng W, Tang Y, Wang H, Tian Z, Bu F, Chen L. Genetic variation in patent foramen ovale: a case-control genome-wide association study. Front Genet. 2025 Jan 13;15:1523304. doi: 10.3389/fgene.2024.1523304. eCollection 2024. PMID 39872005
- [Background] Elliott GC, Gurtu R, McCollum C, Newman WG, Wang T. Foramen ovale closure is a process of endothelial-to-mesenchymal transition leading to fibrosis. PLoS One. 2014 Sep 12;9(9):e107175. doi: 10.1371/journal.pone.0107175. eCollection 2014. PMID 25215881
- [Background] Chabriat H, Joutel A, Dichgans M, Tournier-Lasserve E, Bousser MG. Cadasil. Lancet Neurol. 2009 Jul;8(7):643-53. doi: 10.1016/S1474-4422(09)70127-9. PMID 19539236